CLINICAL TRIAL: NCT04534634
Title: An Open-label, Phase 2, Single-Center Study to Assess the Efficacy and Safety of Interferon-α Combined With Chimeric Antigen Receptor (CAR) T-cell Therapy in Patients With Relapsed and Refractory Acute Lymphoblastic Leukemia（R/R-ALL)
Brief Title: Study of IFN-α Combined With CAR-T Cell Therapy in Relapsed and Refractory Acute Lymphoblastic Leukemia（R/R-ALL）
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Xiaowen Tang, Chief Physician, The First Affiliated Hospital of Soochow University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFN-α+CAR-T
Record Dates: First submitted 2020-08-25; First posted 2020-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: B-cell Acute Lymphoblastic Leukemia
Keywords: IFN-α, CAR-T
MeSH Terms: conditions — Burkitt Lymphoma | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): IFN-α combined with CAR T-cells therapy
  Interventions: Combination Product: IFN-α combined with CAR-T cell therapy
- Control group (No Intervention): CAR T-cells therapy

INTERVENTIONS:
Combination Product: IFN-α combined with CAR-T cell therapy — Adults: 14 daily intramuscular injections 300 million IU of Interferon-α for a 28-day cycle.
  Children: 14 daily intramuscular injections 200mg/m^2 of Interferon-α for a 28-day cycle.
  CAR T cell: (1-2)×10^7/kg, intravenously infusion.
  Other Names: CAR-T cell therapy
  Arms: Experimental group

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of IFN-α combined with CAR-T cell therapy in relapsed and refractory acute lymphoblastic leukemia (R/R ALL).

DETAILED DESCRIPTION:
This is a phase 2, single-center study. The patients will receive IFN-α combined with infusion of CAR T-cells in R/R B-ALL patients. The study participation will be 5 years including treatment and follow-up periods.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed refractory and relapsed acute B-lymphoblastic leukemia.
2. Age 12-65.
3. Eastern Cooperative Oncology Group (ECOG) score 0-2.
4. Target on leukemia is >20% positive detected with flowcytometry.
5. Patients with left ventricular ejection fraction ≥ 0.5 by echocardiography or grade I/II cardiovascular dysfunction according to the New York Heart Association Classification.

5.Patients with aspartate aminotransferase or glutamic-pyruvic transaminase > 3x upper limit of normal or bilirubin > 2.0 mg/dL.

6.No other immunotherapy was received within 3 months.

Exclusion Criteria:

1. Patients are pregnant or lactating.
2. Patients with congenital immunodeficiency.
3. Patients with central nervous system leukemia.
4. Patients with uncontrolled active infection.
5. Patients with active hepatitis B or hepatitis C infection.
6. Patients with HIV infection.
7. Patients with atrial or venous thrombosis or embolism.
8. Patients with myo-infarction or severe arrythmia in the recent 6 months.
9. Other comorbidities that investigators considered not suitable for this study.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 2 years
  ORR includes CR, CRi, MLFS and PR. Complete remission (CR)：Bone marrow blasts <5%; absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count >1.0x 10^9/L; platelet count >100x10^9/L. CR with incomplete hematologic recovery (CRi)：All CR criteria except for residual neutropenia (<1.0x10^9/L) or thrombocytopenia (<100x10^9/L). Morphologic leukemia-free state (MLFS): Bone marrow blasts <5%; absence of blasts with Auer rods; absence of extramedullary disease; no hematologic recovery required. Partial remission (PR): All hematologic criteria of CR; decrease of bone marrow blast percentage to 5% to 25%; and decrease of pretreatment bone marrow blast percentage by at least 50%.

SECONDARY OUTCOMES:
Overall survival (OS) | 2 years
  time from enrollment to the date of death from any cause
Leukemia-free survival (LFS) | 2 years
  time from enrollment to the date of primary refractory disease, or relapse from CR, or death from any cause
Cumulative incidence of relapse(CIR) | 2 years
  time from the date of achievement of a remission until the date of relapse
the duration of CAR-T cells in patients | 2 years
  the time of CAR-T cells' persistence in blood and the copies of CAR-T cells
Number of adverse events | 2 years
  adverse events are evaluated with CTCAE V5.0

CONTACTS AND LOCATIONS:
Overall Officials: xiaowen tang, Ph.D, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China